CLINICAL TRIAL: NCT05846542
Title: Effects of Video-game Based Therapy on Upper Extremity Selective Motor Control and Proprioception in Cerebral Palsy
Brief Title: Video-game Based Therapy in Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gaziantep Islam Science and Technology University (Other)
Responsible Party: Principal Investigator, Demet GÖZAÇAN KARABULUT, Assistant Professor, Gaziantep Islam Science and Technology University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GIBTU-FTR-DGK-3
Record Dates: First submitted 2023-04-24; First posted 2023-05-06 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Cerebral Palsy
Keywords: Cerebral palsy; Virtual reality; Video games; Upper extremity; Rehabilitation
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Video-game based therapy group (Experimental): The video-game based therapy group will receive a conventional physiotherapy and video-game based therapy, two days a week for a total of 8 weeks (15 minutes conventional physiotherapy session+30 minutes video-game based therapy).
  Interventions: Other: Video-game based therapy; Other: Conventional physiotherapy
- Conventional physiotherapy group (Active Comparator): The conventional physiotherapy group individuals will be given a conventional physiotherapy two days per week for a total of 8 weeks (conventional physiotherapy session will last 45 minutes).
  Interventions: Other: Conventional physiotherapy

INTERVENTIONS:
Other: Video-game based therapy — Video-game based therapy will be designed for the individual basis for the upper extremity.
  Arms: Video-game based therapy group
Other: Conventional physiotherapy — Conventional physiotherapy within a specific program

SUMMARY:
The video-based therapy applications; will be applied in a non-three-dimensional (with desktop screen) way. In this application, there are different types of exercise programs that will work the upper extremity movements. The video-based therapy applications will be applied to individuals with Cerebral Palsy (CP) who will be included in the study with the Xbox Kinect 3600 (Microsoft, Washington, USA) device.

This study was planned to examine the effect of video-based therapy on upper extremity selective motor control and proprioception in individuals with Cerebral Palsy.

DETAILED DESCRIPTION:
Spastic CP will be participate the study between the ages of 4 and 18 years. Children's classified with GMFCS and MACS. The eligible participants will be allocated two groups, including video-game based therapy group and conventional physiotherapy control group. All the assessments will be performed before and after the therapy in the 8-week therapy groups.The control group individuals will be given a conventional physiotherapy two days per week for a total of 8 weeks (conventional physiotherapy session will last 45 minutes). The video-game based therapy group will receive a conventional physiotherapy and video-game based therapy, two days a week for a total of 8 weeks (15 minutes conventional physiotherapy session+30 minutes video-game based therapy). All sessions will be performed in the clinic with the specialist physiotherapist.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Cerebral Palsy voluntary participation,
* Age between 4-18 years
* GMFCS Level I-II-III
* MACS Level I-II-III

Exclusion Criteria:

* Not voluntary to participate in the research,
* Botox in the last 6 months,
* Upper limb or spine surgeries in the last 6 months

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2023-04-25 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2023-10-15 (Actual)

PRIMARY OUTCOMES:
Gross Motor Function Classification System (GMFCS) | At Baseline
  Assessing functional level and motor function. Gross motor functions of children with CP are classified in five levels with GMFCS. This is a classification system based on the child's self-initiated movements with emphasis on sitting, displacement and mobility.
Manuel ability classification system (MACS) | At Baseline
  This is a classification system based on the grasping and releasing objects in daily life, and how they use their hands while holding objects. It is classify the hand skills of children with CP between the ages of 4-18.Children with CP are classified in five levels with MACS. The higher level indicates worse hand function
Change from Baseline ABILHAND-Kids at 8 weeks | Change from Baseline at 8 weeks
  Abilhand Kids evaluates manual ability in children with upper extremity disorders. It consists of 21 items and confirmed in CP. The lowest score that can be obtained from the scale is 0 and the highest score is 42. It can be stated that higher scores correspond to more difficulty in activities.
Change from Baseline Selective Control of the Upper Extremity Scale (SCUES) at 8 weeks | Change from Baseline at 8 weeks
  It is a practical and useful assessment tool developed to evaluate upper extremity selective motor control. The administration of the SCUES required patients to perform specific isolated movement patterns at various levels including: shoulder (abduction/adduction); elbow (flexion/extension); forearm (supination/pronation); wrist (flexion/extension); and fingers/thumb (grasp/release). The total score of the SCUES ranges between 0 and 15 and higher scores indicate better selective motor control.
Change from Baseline Clinometer at 8 weeks | Change from Baseline at 8 weeks
  Caliper clinometer (App Development) is a phone application used to measure angle changes in the relevant region. In the evaluation of shoulder and elbow proprioception change will be evaluated.
Change from Baseline Entertainment Scale at 8 weeks | Change from Baseline at 8 weeks
  The entertainment level of sessions and therapy training for individuals will be evaluated with a 0-10 point numerical rating scale (entertainment scale). There are numbers from 0 to 10 on the horizontal line of 10 cm. 0 "Not fun" on the line in the scale; 10 represents "a lot of fun". Entertainment rating will be recorded numerically from 0 to 10.

CONTACTS AND LOCATIONS:
Overall Officials: Demet Gözaçan Karabulut, Study Director — Gaziantep Islam Science and Technology University
Locations (1):
- Demet Gözaçan Karabulut, Gaziantep, None Selected, Turkey (Türkiye)